CLINICAL TRIAL: NCT00655265
Title: A Phase 4 Randomised, Double-Blind, Placebo-Controlled, Parallel-Group, MultiCentre Study of Colesevelam as Add-on Therapy in Patients With Familial Hypercholesterolaemia
Brief Title: A Study of the Safety and Efficacy of Patients With Familial Hypercholesterolaemia Taking Colesevelam as add-on Therapy to Their Existing Medication
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHOL00107; EudraCT 2007-000582-37 (Registry Identifier: EudraCT)
Record Dates: First submitted 2008-04-03; First posted 2008-04-09 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-02

CONDITIONS: Familial Hypercholesterolemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II | interventions — Colesevelam Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Colesevelam hydrochloride film-coated tablets (Experimental)
  Interventions: Drug: Colesevelam hydrochloride film-coated tablets
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colesevelam hydrochloride film-coated tablets — tablets
  Other Names: Cholestagel
  Arms: Colesevelam hydrochloride film-coated tablets
Drug: Placebo — Tablets
  Arms: Placebo

SUMMARY:
This study is designed to assess whether colesevelam given as third line treatment added to a maximal tolerated and stable dose of a statin and ezetimibe is able to further decrease the level of LDL cholesterol in a safe and efficient manner in difficult to treat Familial Hypercholesterolaemia patients who are not at their target level of LDL cholesterol.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a clinical diagnosis of Familial Hypercholesterolaemia defined as EITHER a.Presence of a documented LDL-receptor mutation OR b. History of untreated LDL-cholesterol level above the 95th percentile for sex and age in combination with documentation of at least one of the following: i.Presence of typical tendon xanthomas in the patient or first degree relative. ii. An LDL-cholesterol level above the 95th percentile for age and sex in a first degree relative. iii. Proven coronary artery disease in the patient or in a first degree relative under the age of 60.
* Patients must have provided and undergone lifestyle changes for more than 6 months at the time of Screening
* Patients must have been treated for at least 3 consecutive months preceding the Screening visit with a lipid lowering treatment regimen consisting of maximal tolerated combination of a statin with ezetimibe and are still above their target for LDL cholesterol being 2.5 mmol/L (100 mg/dL)
* Patients must be committed to following the protocol requirements as evidence by written informed consent
* Patients should be comfortable with swallowing 3 placebo tablets

Exclusion Criteria:

* Patients with a known allergy to any of the components used in colesevelam or placebo or any other medications like statin or ezetimibe required for participation in this study
* Patients with a bowel or biliary obstruction
* Patients with secondary causes of hypercholesterolaemia, e.g., dysproteinaemia, hypothyroidism, nephrotic syndrome (defined as proteinuria >2 g/L), obstructive liver disease, other pharmacological therapies, alcoholism
* Patients with triglyceride level of > 3.4 mmol/L
* Patients with dysphagia, swallowing disorders, severe gastrointestinal motility disorders, inflammatory bowel disease, or major gastrointestinal tract surgery
* Patients have undergone LDL-apheresis within one year prior to the screening visit and/or need to undergo LDL-apheresis
* Patients with active liver disease or unexplained persistent elevations in transaminases
* Patients on fenofibrates or on concomitant cholestyramine as this will affect the area under the curve (AUC) of ezetimibe
* Patients with poorly-controlled diabetes (i.e., HbA1c>9% at Screening)
* Patients with clinically significant (CS) abnormal haematology, renal, or other laboratory parameters that could be the result of an underlying malignancy or systemic infection as judged by the investigator
* Patients with a heart transplant, concurrent congestive heart failure (NYHA Class 3 or 4), life-threatening ventricular arrhythmias, unstable angina, recent myocardial infarction within the past 6 months prior to screening, or patients undergoing haemodialysis, or with active disease who may not be healthy enough to successfully complete all protocol requirements
* Fertile women who are pregnant, nursing or using either no or an inadequate form of contraception taking into account the recommendations for adequate intake of oral contraceptives as outlined in concomitant medication section
* Patients with a recent history of alcoholism or drug abuse, or sever emotional behavioural or psychiatric problems who may not be able to adequately comply with the requirements of the study or who may be unable to consent
* Patients receiving experimental medications or participating in another study using an experimental drug or procedure within 30 days prior to signing informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2007-08; Primary Completion 2008-12 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Relative reduction in LDL cholesterol | Between baseline and 6 weeks DB treatment

SECONDARY OUTCOMES:
Relative reduction in HDL, total cholesterol, ApoA1,ApoB,ApoB/ApoA1ratio, triglycerides | Between Baseline and week 6 and week 12 DB treatment
Relative reduction in LDL cholesterol | Between Baseline and week 12 DB treatment

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (8):
- Service d'Endocrinologie, Metabolisme Prevention des Maladies Cardio-Vasculaires, Paris, France
- Kardiologie, Marburg, Germany
- Netherlands (4):
  - Academic Medical Centre, Amsterdam
  - University Medical Centre, Nijmegen
  - University Medical Centre, Utrecht
  - TweeSteden Ziekenhius, Waalwijk
- Centre for Metabolism and Endocrinology, Huddinge, Sweden
- Department of Medicine, University of Manchester, Manchester, United Kingdom